CLINICAL TRIAL: NCT06000293
Title: The Effectiveness of Strengthened Anticipatory Guidance Used in the Ministry of Health Malaysia Infant Oral Health Care Programme: A Cluster Randomised Control Trial
Brief Title: Effectiveness of Strengthened Anticipatory Guidance Used in the MOH Malaysia Infant Oral Health Care Programme
Acronym: MOH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Munalizaini binti Mukhtar, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: USM/JEPeM/KK/23020194; NMRR ID-23-00845-JXN (IIR) (Other: Medical Research & Ethics Committee (MREC) MOH Malaysia)
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Early Childhood Caries; Knowledge, Attitudes, Practice
Keywords: Early Childhood Caries; Knowledge; Practice
MeSH Terms: conditions — Behavior | interventions — Health Education, Dental

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): At baseline, the eligible infant aged 6 months old will undergo clinical oral examination and their primary caregivers will be given the pre-evaluation questionnaires for 6-9 months old. The primary caregivers will then be given the strengthened MOH AG intervention for 6-9 months old infants.
  Following three months, at evaluation 1, the 9-month-old infant will undergo a clinical oral examination, and their primary caregivers will be given the post-evaluation questionnaires for 6-9 months old and pre-evaluation questionnaires for 9-12 months old. The primary caregivers will then be given the strengthened MOH AG intervention for 9-12 months old infants.
  After three months, at evaluation 2, the 12-month-old infant will undergo a clinical oral examination, and their primary caregivers will be given the post-evaluation questionnaires for 9-12 months old.
  Interventions: Other: Oral health education
- Control Group (No Intervention): At baseline, the eligible infant aged 6 months old will undergo clinical oral examination and their primary caregivers will be given the pre-evaluation questionnaires for 6-9 months old. The primary caregivers will be allowed to receive the conventional MOH AG given by oral healthcare providers from the nearest dental clinic.
  Following three months, at evaluation 1, the 9-month-old infant will undergo a clinical oral examination, and their primary caregivers will be given the post-evaluation questionnaires for 6-9 months old and pre-evaluation questionnaires for 9-12 months old.
  After three months, at evaluation 2, the 12-month-old infant will undergo a clinical oral examination, and their primary caregivers will be given the post-evaluation questionnaires for 9-12 months old.

INTERVENTIONS:
Other: Oral health education — Anticipatory Guidance (AG) provided to the primary caregivers-infant pairs in the intervention group
  Other Names: Dental health education
  Arms: Treatment Group

SUMMARY:
This study aimed to assess the effectiveness of strengthened anticipatory guidance (AG) used in MOH Malaysia Infant Oral Healthcare Programme in preventing early childhood caries (ECC) lesions and improving caries risk of infants in Negeri Sembilan and their primary caregiver's knowledge and practice on infant oral healthcare

DETAILED DESCRIPTION:
This randomised control trial study will be conducted at six government Maternal and Child Health Clinics (MCHCs) in Negeri Sembilan District, Malaysia. The samples comprised of 220 primary caregivers-infant pairs (110 pairs in the intervention group, and 110 pairs in the control group). A strengthened infant oral health module named the Oral Health Infant Module Anticipatory Guidance (OHIM AG) was designed to provide anticipatory guidance to the intervention group at three-month intervals over 6 months. The control group will receive the conventional Ministry of Health Anticipatory Guidance (MOH AG). The effectiveness of OHIM AG on early signs of childhood caries lesions development, caries risk of infants, and primary caregivers's knowledge and practice on infant oral healthcare will be assessed after six months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* The infant and primary caregivers (parents/ caregivers) are a Malaysian citizen
* Primary caregivers can read and understand Bahasa Malaysia. This is because the AG will be conducted in Bahasa Malaysia, and the questionnaires are also in Bahasa Malaysia.

Exclusion Criteria:

* Infants with special needs, chronic diseases or conditions (e.g., stunting, failure to thrive and low birth weight) who are at risk for oral problems (e.g., higher risk of caries due to presence of hypomineralisation and hyperplasia) and require special oral health care.

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Early dental caries lesion and dental caries risk exposure among infants | 6 months
  The prevalence of early dental caries lesion and dental caries risk exposure between infants in the intervention and control groups.
Knowledge and practice score on infant oral health care among primary caregivers (parents/ caregivers) | 6 months
  The knowledge and practice score on infant oral health care between primary caregivers in the intervention and control groups.
  The response options for knowledge items are true, false and don't know. A score of 1 will be given to correct answers and a score of 0 for incorrect and don't know answers. A higher score indicates better knowledge.
  Each practice item is given 4 response options, including a never. The remaining three responses will include one correct or appropriate practice and two incorrect or inappropriate responses. A score of 1 will be given for the correct or appropriate answers, and a score of 0 will be given for inaccurate or inappropriate and never answers. A higher score indicates better practice.
  In addition to individual domain scores, an overall score for knowledge and practice on infant oral health care can be determined by dividing the summed score from knowledge and practice domains by the total possible score.

CONTACTS AND LOCATIONS:
Overall Officials: Munalizaini Mukhtar, Principal Investigator — Universiti Sains Malaysia

IPD SHARING:
Plan to Share IPD: No
Data obtained from this study will be published for knowledge purposes and will be presented as grouped data and thus will not identify the respondents individually. The data of subjects will be kept private and confidential for up to about five years after this study is completed and will be destroyed. Subjects can write to the investigators to request access to study findings. The data will not be disclosed to any parties working on this project unrelated to this study.